CLINICAL TRIAL: NCT06848478
Title: Level Up! (The Combined and Independent Effects of Exercise Training and Dietary Enhancement on Cardiometabolic Health in Adolescents With Obesity)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 287133; USDA/ARS 6026-10700-001-000D (Other Grant/Funding Number: United States Department of Agriculture (USDA) - Agricultural Research Service (ARS))
Record Dates: First submitted 2025-01-17; First posted 2025-02-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: exercise; obesity; diet; cardiometabolic
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants receive the standard of care for treating Class I and II obesity.
- Exercise intervention (Experimental): In addition to the standard of care, participants engage in exercise coaching and a 12-week exercise program, encompassing three 60-minute supervised sessions per week.
  Interventions: Behavioral: Exercise Intervention
- Nutritional Intervention (Experimental): In addition to the standard of care, participants receive dietary coaching and engage in a 12-week daily dietary program enriched with a blend of fruits and vegetables.
  Interventions: Behavioral: Nutritional Intervention
- Exercise and Nutritional Intervention (Experimental): In addition to the standard of care, participants receive a combined exercise and dietary intervention, as described in the other two intervention arms.
  Interventions: Behavioral: Exercise Intervention; Behavioral: Nutritional Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — In addition to the standard of care, participants engage in exercise coaching and a 12-week exercise program, encompassing three 60-minute supervised sessions per week.
  Arms: Exercise and Nutritional Intervention; Exercise intervention
Behavioral: Nutritional Intervention — In addition to the standard of care, participants receive dietary coaching and engage in a 12-week daily dietary program enriched with a blend of fruits and vegetables.
  Arms: Exercise and Nutritional Intervention; Nutritional Intervention

SUMMARY:
The goal of this clinical trial is to learn how exercise and diet quality affect the health of adolescents with obesity. The main questions it aims to answer are:

* Does exercise improve cardiometabolic health in adolescents with obesity?
* Does enriching the diet with fruits and vegetables improve cardiometabolic health in adolescents with obesity?
* Do exercise and a fruit and vegetable diet together provide greater health benefits than either one alone in adolescents with obesity?

Researchers will compare four groups to see how exercise and diet impact health:

* Standard Care Group: Receives the usual care for obesity.
* Exercise Group: Receives weekly exercise coaching and participates in a 12-week exercise program.
* Diet Group: Receives weekly dietary coaching and eats a diet enriched with fruits and vegetables for 12 weeks.
* Combined Exercise and Diet Group: Receives both exercise and dietary programs, namely weekly exercise and dietary coaching, participation in a 12-week exercise program, and daily consumption of fruits and vegetables for 12 weeks.

During the 12-week study, participants will attend three study visits to:

* Provide blood, stool, and urine samples.
* Answer questions about health, sleep, diet, and physical activity.
* Undergo body scans to measure fat, lean, and bone mass.
* Complete blood vessel function and liver fat content assessments.
* Assess resting exergy expenditure.
* Complete fitness tests.
* Wear a fitness tracker to monitor physical activity and sleep patterns.

DETAILED DESCRIPTION:
The Level Up! study is a 12-week randomized controlled trial designed to investigate the independent and combined effects of exercise training and dietary enrichment on cardiometabolic health in adolescents with obesity. The study will enroll adolescents participating in an obesity treatment program. Participants will be randomly assigned to one of four groups: standard of care, exercise, dietary, or combined exercise and dietary intervention.

Each participant will attend three assessment visits at baseline, week 6, and week 12 at the Arkansas Children's Nutrition Center (ACNC). The following key measurements will be conducted:

* Body Composition: Dual-Energy X-ray Absorptiometry (DXA)
* Metabolic Profile: Fasting blood markers, including glucose, lipid profile, and insulin resistance
* Vascular Function: Brachial artery flow-mediated dilation (ultrasound)
* Liver Fat Content: Elastography
* Continuous Glucose Monitoring: Interstitial sensor-based glucose measurement
* Resting Metabolic Rate: Indirect calorimetry
* Aerobic Capacity: Cardiopulmonary exercise test (spirometry)
* Muscle Strength: Dynamometry
* Physical Activity & Sleep: Accelerometry
* Dietary Intake: 3-day food records

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 13 to 17 years.
* Newly enrolled in a weight management program.
* Excessive weight: Class I obesity I (≥95% percentile to < 120% of the 95th percentile), class II Obesity (≥120 to <140% of the 95th percentile, or BMI ≥35 to < 40 g/m2).
* Less than 60 min/day of moderate to vigorous physical activity.
* Fruit intake ≤ 1.5 cup equivalent per day.
* Vegetable intake ≤ 1.5 cup equivalent per day.
* Medical release.

Exclusion Criteria:

* Type 2 diabetes mellitus.
* Asthma that requires daily use of inhalers to keep symptoms under control.
* Asthma that requires the use of rescue inhalers (e.g., albuterol) >2 days per week
* Exercise-induced asthma.
* Autism spectrum disorder (e.g., Autistic disorder, Rett disorder, Asperger disorder, childhood disintegrative disorder, pervasive developmental disorder not otherwise specified (PDD-NOS).
* Epilepsy.
* Cancer.
* Chronic kidney disease.
* Hormonal disease (e.g., hypothyroidism and growth hormone deficiency).
* Autoimmune diseases (e.g., lupus, thyroiditis, juvenile idiopathic arthritis).
* Bleeding disorders (e.g., hemophilia).
* Chronic infections (e.g., HIV, hepatitis B, hepatitis C).
* Other pre-existing medical conditions or medications as determined by the investigators to affect the outcomes of interest.
* Pregnancy.
* Dislike of > 1 study product assessed at the initial visit.
* Parent/child refusal to have blood drawn.
* Refusal to authorize study investigators to access data from the clinical records.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-10-27 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Group differences in composite score of cardiometabolic health changes over time. | Baseline, 6 weeks, and 12 weeks.
  The primary outcome is a composite score of cardiometabolic health status. The score is calculated as the mean of specific z-scores for the following markers: fasting triglycerides (mg/dL), total cholesterol/HDL-cholesterol ratio, HOMA2-IR, systolic blood pressure (mmHg), fat-mass-index [whole-body fat mass (kg)/height² (m²)], and inverse peak oxygen uptake (mL O₂/kg/min). The composite score is computed as the mean of the standardized z-scores for each marker, providing an overall measure of cardiometabolic health status.

SECONDARY OUTCOMES:
Group differences in low-density lipoprotein (LDL) cholesterol (mg/dL) changes over time. | Baseline, 6 weeks, and 12 weeks.
Group differences in fow-mediated dilation (%) changes over time. | Baseline, 6 weeks, and 12 weeks.
Group differences in liver steatosis (dB/m) changes over time. | Baseline and 12 weeks.
Group differences in appendicular lean mass index changes over time. | Baseline, 6 weeks, and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Borsheim, Ph.D, Principal Investigator — Arkansas Children's Research Institute
Locations (2):
- United States (2):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Arkansas Children's Nutrition Center, Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: Undecided